CLINICAL TRIAL: NCT00810784
Title: Evaluation of Venous Thromboembolism (VTE) Prophylaxis in Medically Ill Patients
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Robert Pendleton, M.D., Associate Professor, University of Utah, University of Utah
Other Study IDs: UUHSC-IRB-00018164
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism; Prevention; Quality Improvement; Education; Compliance with VTE prophylaxis
MeSH Terms: conditions — Venous Thromboembolism | interventions — Educational Status

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients cared for before our intervention.
- 2: Patients cared for after our intervention.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — (1) a risk-assessment tool completed at the time of a hospital admission, (2) structured educational sessions on VTE prevention, and (3) audit-feedback where institutional data was reviewed during the educational sessions. These sessions were given once to the clinical pharmacists and on three separate occasions to the medicine house officers.
  Groups: 2

SUMMARY:
VTE prophylaxis is not as routinely employed in medically ill patients as compared to surgical patients. This retrospective chart review project will evaluate the effectiveness of VTE prophylaxis in medically ill patients at the University of Utah Hospitals and Clinics compared to current literature. The study will ultimately serve as a quality improvement project to help improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at the University of Utah on one our medical services.

Exclusion Criteria:

* Patients received therapeutic anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data was collected on consecutive patients ≥18 years with a hospital length of stay of >48 hours admitted to the cardiology, pulmonary, or general medical services. Admission dates were a sample of two different two-week blocks (January 1-14, 2006 and April 1-14, 2006). These blocks were chosen to be consistent with dates of analysis in the pre-intervention cohort. Patients receiving therapeutic anticoagulation were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2005-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rondina, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Stinnett JM, Pendleton R, Skordos L, Wheeler M, Rodgers GM. Venous thromboembolism prophylaxis in medically ill patients and the development of strategies to improve prophylaxis rates. Am J Hematol. 2005 Mar;78(3):167-72. doi: 10.1002/ajh.20281. PMID 15726600